CLINICAL TRIAL: NCT05619432
Title: VRision Program - Scaling of a Validated Virtual Reality Training Program for Improving Vision in Older Adults
Brief Title: Re:Garde Program - Training and Maintaining Visual Perception in Older Adults
Acronym: Re:Garde
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: University Health Network, Toronto (Other)
Collaborators: Perley Rideau (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-5847
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Vision, Low; Visual Impairment
MeSH Terms: conditions — Vision, Low; Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Clinic Setting (Experimental): Participants will complete their virtual reality (VR) visual training program by visiting a local clinic and using the head-mounted display (HMD) provided. Participants will receive initial training on using the device and software and are expected to complete their 6-weeks of visual training independently at the clinic. Additional training and FAQ materials will be available on site for participants to use as reference.
  Interventions: Device: HMD: Immersive VR
- Group B: Home Setting (Experimental): Participants will complete their virtual reality (VR) visual training program from their own homes using a head-mounted display (HMD) that is on loan for the study. Participants will receive initial training on using the device and software at the clinic and will take home the HMD to complete their 6-weeks of visual training independently from home. Additional training and FAQ materials will be given to participants to use as reference.
  Interventions: Device: HMD: Immersive VR

INTERVENTIONS:
Device: HMD: Immersive VR — The device application involves the 3D multiple-object-tracking (3D-MOT) paradigm composed of 8 high-contrast spheres which are adapted to the visual ability of participant (luminosity and size). The initial speed of the spheres is adjustable and determined during the inclusion visit.
  STIMULATION:
  One or more of the spheres is temporarily cued (target). Then all spheres move for 20 seconds following random linear paths, bouncing on one another and on the walls of a virtual 3D cube when collisions occur. After 20 seconds, the movement stops and the participant is asked to select, using a laser pointer, the initially cued target(s) among the eight spheres. If the selection is correct the speed of the spheres in the next trial is increased. If the selection is incorrect the speed of the spheres in the next trial is decreased.
  Based on performance, stimulations will be adjusted to change difficulty level (e.g. changing backgrounds, number of cued balls, etc.)

SUMMARY:
Seniors deal with considerable visual demands (driving, communicating, traveling) and reduced vision affects their quality of life, ability to enjoy activities, and age-in-place. Vision loss has a heavy, increasing, economical and social burden. It can also have substantial impacts on caregivers physically, psychologically, and financially because one tends to miss more work, be less productive, and thus have fewer job opportunities.

This registration will describe the clinical portion of a larger study designed to evaluate both the feasibility and effectiveness of the Re:Garde Program, a Virtual Reality (VR) visual training program for older adults to help maintain visual perception to promote quality of life and prolonged independence. In partnership with our care partners the investigators will implement the Re:Garde Program at an interprofessional clinic and as part of a loaning program for older adults to use in the home.

The clinical portion of this study will look at how effective the Re:Garde program is at maintaining or improving visual perception, ability to conduct activities of daily living (e.g. read, drive, cook, exercise etc.), general wellness, and quality of life. The feasibility of implementing this program in the two settings will be evaluated separately as part of the full protocol.

DETAILED DESCRIPTION:
This will be an interventional, pragmatic, pilot study with a target total recruitment of 30 participants (15 per arm). The study duration is 7 weeks. Participants will be assigned to one of two arms: Clinic Setting vs Home Setting.

SCREENING & BASELINE TEST

At the initial visit in the clinic, participants will be screened for exclusion criteria and practice a condensed version of the immersive VR (IVR) stimulation using the head-mounted display (HMD). Following stimulation participants will be assessed for IVR sensitivity, or cybersickness, using the Virtual-Reality Induced Symptoms and Effects (VRISE) questionnaire. Finally participants will be asked to complete vision tests within the VR headset (for visual attention and cognition) and a series of questionnaires corresponding to visual perception, ability to perform activities of daily living, and quality of life. Participants in the home-arm will take home an HMD along with a package of questionnaires for the duration of the study.

INTERVENTION

Participants of the study will perform their visual training on the HMD every other day for six weeks (21 sessions total). The clinic-arm participants will train at the clinic using the HMD provided. The home-arm participants will train using the HMD on loan to them for the duration of the study.

Each training session (to be completed every other day) will contain three blocks of 15 audiovisual stimulation tasks. Each task lasts for 20 seconds of audiovisual IVR stimulation (3D-Multi Object Tracking + correlated sound). There will be a 2-min break between each of the three blocks of tasks. After each session, the participant will answer the VRISE questionnaire through the HMD. Data from the IVR stimulation and the VRISE score will be sent automatically through Wi-Fi in real-time to a dedicated and secured laboratory computer located at Krembil Research Institute after each session. The total time for the training session should be approximately 15 minutes.

At the mid-point of intervention (end of week 3) participants will repeat the visual tests and questionnaires from baseline.

POST-INTERVENTION

After participants complete their 6-week intervention program they will repeat the visual tests and questionnaires from baseline along with a new questionnaire to evaluate the quality of the VR software in terms of user experience. Subjects participating in the loaning program will schedule a home visit where the VR equipment and questionnaires will be collected at this point. All participants will also be interviewed to collect feedback on their experience with the device, feasibility of the therapy, and overall experience.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* Have self-reported healthy vision or only self-reported vision issues
* Can have corrected vision and use glasses/contacts with the VR headset
* Have access to Wi-Fi if participating from home

Exclusion Criteria:

* Vision impairments (such as glaucoma, macular degeneration, etc.) as diagnosed by a medical professional
* Cervical conditions, injuries, or open face wounds that would make it unsafe to use the VR headset
* Cannot speak or understand English

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in self-reported vision based on the Activities of Daily Vision Scale (ADVS) | Initial Visit (Day 1), Mid-point (end of Week 3), Treatment completion (Week 7)
  This 19-item questionnaire will ask participants about a series of daily activities that some individuals with visual problems find challenging to perform. These activities are categorized into five subscales (distance vision, near vision, glare disability, night driving, and daytime driving). Each subscale is scored between 0 (inability to perform the activity because of visual difficulty) and 100 (no visual difficulty).
Changes from baseline in self-reported independence/autonomy using the Instrumental Activities of Daily Living (IADL) Scale | Initial Visit (Day 1), Mid-point (end of Week 3), Treatment completion (Week 7)
  This questionnaire will ask participants to rate their degree of independence for eight (8) different common activities of daily living (e.g. food preparation, handling own medication, etc.) The summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women and 0 through 5 for men to avoid potential gender bias.
Changes from baseline in self-reported well-being using the World Health Organization-5 Well-Being Index (WHO-5) | Initial Visit (Day 1), Mid-point (end of Week 3), Treatment completion (Week 7)
  This questionnaire for general mental well-being consists of five (5) statements and will ask participants to rate how often they have agreed with each statement in the past two weeks. The raw score ranges from 0 (worst possible quality of life) to 25 (best possible quality of life).
Changes from baseline in visual attention and speed using Re:ViewD | Initial Visit (Day 1), Mid-point (end of Week 3), Treatment completion (Week 7)
  This vision test will be completed within the VR headset and will measure visual processing speed, sustained visual attention, and divided visual attention. This is a VR version of the Useful Field of View (UFoV) test which has been extensively used to measure visual attention in healthy individuals and older adults with low vision.
Changes from baseline in visual cognition using Re:ShapeD | Initial Visit (Day 1), Mid-point (end of Week 3), Treatment completion (Week 7)
  This vision test will be completed within the VR headset and will measure visual cognition. This is a VR version of the Motor-Free Visual Perception Test (MVPT) which evaluates visual perception, in particular discrimination, figure-ground, visual memory, spatial relationships, and visual closure.
Virtual-Reality Induced Symptoms and Effects (VRISE) - initial screening | Initial Visit (Day 1)
  This questionnaire is made up of five (5) questions related to possible cybersickness symptoms and will be completed within the VR headset by using the hand controller. Participants will complete the VRISE immediately after being trained to use Re:Garde at the initial visit. The VRISE score ranges from 5 (very intense level of symptoms and effects) to 35 (very low level of symptom and effects).
Virtual-Reality Induced Symptoms and Effects (VRISE) - intervention period | Every other day with training session (Weeks 1-6)
  This questionnaire is made up of five (5) questions related to possible cybersickness symptoms and will be completed within the VR headset by using the hand controller. Participants will complete the VRISE immediately before and after each VR training session. The VRISE score ranges from 5 (very intense level of symptoms and effects) to 35 (very low level of symptom and effects).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Reber, PhD, Principal Investigator — University Health Network, Toronto; Lora Appel, PhD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Perley Health, Ottawa, Ontario
  - Krembil Research Institute, UHN, Toronto, Ontario

REFERENCES:
- [Background] Graf C. The Lawton instrumental activities of daily living scale. Am J Nurs. 2008 Apr;108(4):52-62; quiz 62-3. doi: 10.1097/01.NAJ.0000314810.46029.74. PMID 18367931
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Mangione CM, Phillips RS, Seddon JM, Lawrence MG, Cook EF, Dailey R, Goldman L. Development of the 'Activities of Daily Vision Scale'. A measure of visual functional status. Med Care. 1992 Dec;30(12):1111-26. doi: 10.1097/00005650-199212000-00004. PMID 1453816
- [Background] Saredakis D, Szpak A, Birckhead B, Keage HAD, Rizzo A, Loetscher T. Factors Associated With Virtual Reality Sickness in Head-Mounted Displays: A Systematic Review and Meta-Analysis. Front Hum Neurosci. 2020 Mar 31;14:96. doi: 10.3389/fnhum.2020.00096. eCollection 2020. PMID 32300295
- [Background] Wittinghofer A, Warren WF, Leberman R. Structural requirements of the GDP binding site of elongation factor Tu. FEBS Lett. 1977 Mar 15;75(1):241-3. doi: 10.1016/0014-5793(77)80095-1. No abstract available. PMID 323049
- [Background] Leat SJ, Lovie-Kitchin J. Visual impairment and the useful field of vision. Ophthalmic Physiol Opt. 2006 Jul;26(4):392-403. doi: 10.1111/j.1475-1313.2006.00383.x. PMID 16792739
- [Background] Richards E, Bennett PJ, Sekuler AB. Age related differences in learning with the useful field of view. Vision Res. 2006 Nov;46(25):4217-31. doi: 10.1016/j.visres.2006.08.011. Epub 2006 Oct 5. PMID 17027061
- [Background] Brown T, Elliott S. Factor structure of the Motor-Free Visual Perception Test-3rd edition (MVPT-3). Can J Occup Ther. 2011 Feb;78(1):26-36. doi: 10.2182/cjot.2011.78.1.4. PMID 21395195